CLINICAL TRIAL: NCT04014816
Title: The Frequency, Risk Factors, and Complications of Gastrointestinal Dysfunction During Enteral Nutrition in Critically Ill Patients
Brief Title: Gastrointestinal Dysfunction During Enteral Nutrition in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Ayancık State Hospital (Other Government)
Responsible Party: Principal Investigator, Ayse Gulsah Atasever, Anesthesiology Specialist, Ayancık State Hospital
Other Study IDs: 2014/1870
Record Dates: First submitted 2019-07-04; First posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Gastrointestinal Disease; Constipation; Intolerance; Nutritional; Diarrhea
Keywords: ICU
MeSH Terms: conditions — Gastrointestinal Diseases; Constipation; Diarrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: Patients who had GI dysfunction (Group I) for one or more occasions.
  Interventions: Other: MDR bacteria positivity; Other: negative fluid balance
- Group II: Patients who had normal GI function (Group II) for one or more occasions.
  Interventions: Other: MDR bacteria positivity; Other: negative fluid balance

INTERVENTIONS:
Other: MDR bacteria positivity — A total of 137 patients who received nasogastric tube feeding in an ICU of a tertiary hospital were enrolled.
Other: negative fluid balance — A total of 137 patients who received nasogastric tube feeding in an ICU of a tertiary hospital were enrolled.

SUMMARY:
Gastrointestinal (GI) motility disorders in intensive care patients remain relatively unexplored. Nowadays, the frequency, risk factors and complications of GI dysfunction during enteral nutrition (EN) become more questionable. Our aim is to evaluate the frequency, risk factors and complications of GI dysfunction during EN in the first 2 weeks of the intensive care unit (ICU) stay and to identify precautions to prevent the development of GI dysfunction and avoid complications.

DETAILED DESCRIPTION:
Critical illness is typically associated with a catabolic stress state in which patients demonstrate a systemic inflammatory response coupled with complications of increased infectious morbidity, multiple organ dysfunction, prolonged hospitalization, and disproportionate mortality. Suspension of feeding and the resultant inability to reach nutritional goals is one complication of gastrointestinal (GI) dysfunction, but there are others (mucosal barrier disruption, altered motility, atrophy of the mucosa, and reduced mass of gut-associated lymphoid tissue) that may explain the greater length of stay (LOS) and death rate with GI dysfunction. In Europe and the United States, nutritional administration guidelines recommend primarily enteral nutrition (EN) for hemodynamically stable intensive care unit (ICU) patients. Providing EN in these patients has been shown to be superior to parenteral nutrition. GI complications such as constipation, delayed gastric emptying, diarrhea, and vomiting may occur in up to 50% of mechanically ventilated patients and adversely affect ICU mortality and LOS. Nevertheless, there is no consensus for obtaining a precise assessment of GI function.Diagnosis of GI dysfunction in ICU patients is complex and relies on clinical symptoms. Lack of validated markers of GI system dysfunction is often misdiagnosed and poorly managed in the ICU. The role of nutrition in critical illness is important, but there is an increasing evidence and broadening consensus that aggressive early feeding as well as prolonged underfeeding both should be avoided. Avoidance of complications like malnutrition, aspiration of gastric contents, wound infections, and decubitus through GI dysfunction is an important part of management of patients with GI failure.

ELIGIBILITY:
Inclusion Criteria:

Older than 18 years old. Stay longer than 48 hours at ICU.

Exclusion Criteria:

Has enterostomy/colostomy or diagnosis of GI bleeding. Prone position. Laxative drug use. Clostridium Difficile infection positivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this prospective observational study, 137 out of 226 patients consecutively admitted into a mixed medical-surgical ICU from 1 January 2015 to 31 June 2015 were enrolled.
Sampling Method: Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2015-07-01 (Actual)

PRIMARY OUTCOMES:
The incidence of GI dysfunction | up to 14 days.
  Constipation, diarrhea, UDI

SECONDARY OUTCOMES:
The sequential organ failure assessment(SOFA) score | at admission.
  SOFA Score is a mortality pre-score that is based on the degree of dysfunction of six organ systems. Each organ system is assigned a point value from 0 (normal)to 4 (high degree of dysfunction/failure). The SOFA score ranges from 0 to 24.The highest SOFA score correlates with highest mortality rates. Scores of more than 11 corresponded to mortality of more than 80%.
Hypoalbuminemia | up to 14 days.
  below 2,5 g/dl
Catecholamine use | up to 14 days.
  mcg
Length of hospital stay | through study completion, which is 6 months time period.
  days

CONTACTS AND LOCATIONS:
Overall Officials: Evren Senturk, Assoc. Prof, Study Director — Koc University Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Atasever AG, Ozcan PE, Kasali K, Abdullah T, Orhun G, Senturk E. The frequency, risk factors, and complications of gastrointestinal dysfunction during enteral nutrition in critically ill patients. Ther Clin Risk Manag. 2018 Feb 23;14:385-391. doi: 10.2147/TCRM.S158492. eCollection 2018. PMID 29503558
- See also: Upper digestive intolerance during enteral nutrition in critically ill patients: frequency, risk factors, and complications. Crit Care Med. 2001;29:1955-1961. — https://www.ncbi.nlm.nih.gov/pubmed/11588461
- See also: Diarrhoea in the ICU: respective contribution of feeding and antibiotics. Crit Care. 2013;17:R153. — https://www.ncbi.nlm.nih.gov/pubmed/23883438
- See also: Enteralnutrition-relatedgastrointestinalcomplicationsin critically ill patients: a multicenter study: The Nutritional and Metabolic Working Group of the Spanish Society of Intensive Care Medicine and Coronary Units. Crit Care Med. 1999;27:1447-1 — https://www.ncbi.nlm.nih.gov/pubmed/10470748